CLINICAL TRIAL: NCT00195065
Title: Cornell Translational Behavioral Science Research Consortium: Asthma Qualitative Study
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Mary E. Charlson, MD, Weill Cornell Medical College
Other Study IDs: N01-HC-25196 (9811003566); N01HC25196 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Asthma
Keywords: Asthma; Behavior change; Physical activity; Risk reduction
MeSH Terms: conditions — Asthma; Motor Activity; Risk Reduction Behavior

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Semi-structured, open-ended interviews

SUMMARY:
To explore and illuminate the cultural, social, and psychological factors that either facilitate or serve as barriers to behavioral change in asthma patients.

DETAILED DESCRIPTION:
1. Through a series of open-ended questions we will explore and build a better understanding of how different patient populations view asthma and the difficulties they face in changing behavior. In addition the responses to such questions should help us to better understand and anticipate some of the barriers and issues that participants may face in successfully changing their behaviors.
2. The second objective is to use the responses obtained to inform how an intervention of positive affect induction and self-affirmation should be operationalized and tailored.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for this study if their physicians consider them medically able to participate, if they are 18 years of age or older, and if they have a diagnosis of mild to moderate asthma based on the NHLBI Asthma Expert Panel's classification system which rates symptoms, frequency of exacerbations, nocturnal attacks, activity restriction, use of medications, and pulmonary function.

Exclusion Criteria:

Patients will be excluded from this study for the following reasons:

* If they are unable to walk several blocks for whatever reason;
* If they have musculoskeletal or neurological deficits that preclude increased physical activity;
* If they have other pulmonary diseases;
* If they have cardiac disease or other severe comorbidity;
* If they are unable to provide informed consent because of cognitive deficits;
* If they refuse to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-04; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Mancuso, MD, Principal Investigator — Weill Medical College of Cornell University; Mary E Charlson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital-Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- [Background] Mancuso CA, Peterson MG. Different methods to assess quality of life from multiple follow-ups in a longitudinal asthma study. J Clin Epidemiol. 2004 Jan;57(1):45-54. doi: 10.1016/S0895-4356(03)00248-8. PMID 15019010
- [Background] Mancuso CA, Rincon M, Robbins L, Charlson ME. Patients' expectations of asthma treatment. J Asthma. 2003 Dec;40(8):873-81. doi: 10.1081/jas-120023578. PMID 14736086
- [Background] Mancuso CA, Rincon M, McCulloch CE, Charlson ME. Self-efficacy, depressive symptoms, and patients' expectations predict outcomes in asthma. Med Care. 2001 Dec;39(12):1326-38. doi: 10.1097/00005650-200112000-00008. PMID 11717574
- [Background] Mancuso CA, Peterson MG, Charlson ME. Effects of depressive symptoms on health-related quality of life in asthma patients. J Gen Intern Med. 2000 May;15(5):301-10. doi: 10.1046/j.1525-1497.2000.07006.x. PMID 10840265
- [Result] Mancuso CA, Sayles W, Robbins L, Phillips EG, Ravenell K, Duffy C, Wenderoth S, Charlson ME. Barriers and facilitators to healthy physical activity in asthma patients. J Asthma. 2006 Mar;43(2):137-43. doi: 10.1080/02770900500498584. PMID 16517430